CLINICAL TRIAL: NCT06051955
Title: Evaluation of an Oral Sodium Sulfate Solution for Patients With Prior Difficult or Incomplete Cleansing, a Progressive Case Series.
Brief Title: Evaluation of an Oral Sodium Sulfate Solution for Patients With Prior Difficult or Incomplete Cleansing
Acronym: OSS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lawrence Charles Hookey (Other)
Collaborators: Pendopharm (Industry)
Responsible Party: Sponsor-Investigator, Lawrence Charles Hookey, Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 6039506
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Colonoscopy; Bowel Preparation
Keywords: Oral sodium sulfate
MeSH Terms: interventions — sodium sulfate

STUDY DESIGN:
Intervention Model Description: This study will enroll participants who have experienced difficult or incomplete bowel cleansing in the past. All participants will use oral sodium sulfate as their cleansing agent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- oral sodium sulfate (Other): OSS is a colon cleansing agent administered in a split dose fashion, inducing diarrhea by drawing water into the intestine.
  Interventions: Other: oral sodium sulfate

INTERVENTIONS:
Other: oral sodium sulfate — All participants enrolled in this study will use Oral Sodium Sulfate as their bowel cleansing agent.

SUMMARY:
This case series aims to evaluate the effectiveness and tolerability of Oral Sulfate Solution (OSS) in patients who had previously experienced poor colonoscopy preparation.

DETAILED DESCRIPTION:
This study aims to evaluate the effectiveness of Oral Sodium Sulfate (OSS) in patients who have had poor colon preparation in the past. The study includes patients who had issues during their previous colonoscopy, such as needing extensive washing, inadequate preparation, a recommendation for shorter surveillance intervals, or adequate preparation for larger polyps but not smaller lesions.

Poor colon cleansing during a colonoscopy can lead to more prolonged procedures, lower polyp detection rates, and the need for repeat procedures with shorter surveillance intervals. OSS is a low-volume osmotic agent that causes diarrhea and colon cleansing by drawing water into the intestine. Health Canada and the FDA have approved it, and it is given in two 177ml bottles in a split dose. OSS is known for its good effect, ease of use, and tolerability, and it may be a better option than traditional cleansing agents.

All participants will receive OSS and instructions for use before their next surveillance colonoscopy. The study will use questionnaires and patient diaries to assess the effectiveness of OSS and patient compliance and tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Patients Age 18 to 80 inclusive
2. Able to read and understand the English language
3. History of poor bowel prep defined as:

   * Required extensive washing, as noted in the narrative of the endoscopist report.
   * Inadequate preparation
   * Endoscopist recommended shorter interval surveillance due to poor prep
   * adequate for polyps >5mm but not smaller lesions

Exclusion Criteria:

1. Patients who have inflammatory bowel disease
2. Patients with ileus or bowel obstruction
3. Patients with history of colorectal resection
4. Patients receiving combined upper and lower endoscopies
5. Patients with ascites
6. Patients with previously documented severe renal impairment
7. Unable to provide consent
8. Pregnant or lactating female (females of child-bearing potential will undergo urine pregnancy testing)
9. Patients who have had a recent myocardial infarction(<6months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Effectiveness | 1-2 days
  The primary outcome is proportion of patients with an adequate preparation (Boston preparation scale 6 or greater, with no section less than 2).

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Hookey, Principal Investigator — Queen's University
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnson DA, Barkun AN, Cohen LB, Dominitz JA, Kaltenbach T, Martel M, Robertson DJ, Boland CR, Giardello FM, Lieberman DA, Levin TR, Rex DK; US Multi-Society Task Force on Colorectal Cancer. Optimizing adequacy of bowel cleansing for colonoscopy: recommendations from the US multi-society task force on colorectal cancer. Gastroenterology. 2014 Oct;147(4):903-24. doi: 10.1053/j.gastro.2014.07.002. No abstract available. PMID 25239068
- [Background] Oldfield EC 4th, Johnson DA, Rex DK. Prescribing Colonoscopy Bowel Preparations: Tips for Maximizing Outcomes. Am J Gastroenterol. 2023 May 1;118(5):761-764. doi: 10.14309/ajg.0000000000002110. Epub 2022 Dec 26. No abstract available. PMID 36573902
- [Background] Wang CN, Yang R, Hookey L. Does It work in Clinical Practice? A Comparison of Colonoscopy Cleansing Effectiveness in Clinical Practice Versus Efficacy from Selected Prospective Trials. J Can Assoc Gastroenterol. 2020 Jun;3(3):111-119. doi: 10.1093/jcag/gwy070. Epub 2019 Feb 12. PMID 32395685
- [Background] Hookey LC, Vanner S. A review of current issues underlying colon cleansing before colonoscopy. Can J Gastroenterol. 2007 Feb;21(2):105-11. doi: 10.1155/2007/634125. PMID 17299615
- [Background] Anastassopoulos K, Farraye FA, Knight T, Colman S, Cleveland MV, Pelham RW. A Comparative Study of Treatment-Emergent Adverse Events Following Use of Common Bowel Preparations Among a Colonoscopy Screening Population: Results from a Post-Marketing Observational Study. Dig Dis Sci. 2016 Oct;61(10):2993-3006. doi: 10.1007/s10620-016-4214-2. Epub 2016 Jun 9. PMID 27278957
- [Background] Rex DK, DiPalma JA, McGowan J, Cleveland Mv. A comparison of oral sulfate solution with sodium picosulfate: magnesium citrate in split doses as bowel preparation for colonoscopy. Gastrointest Endosc. 2014 Dec;80(6):1113-23. doi: 10.1016/j.gie.2014.05.329. Epub 2014 Jul 12. PMID 25028274
- [Background] Yang HJ, Park SK, Kim JH, Im JP, Yeom DH, Seo GS, Park DI. Randomized trial comparing oral sulfate solution with 4-L polyethylene glycol administered in a split dose as preparation for colonoscopy. J Gastroenterol Hepatol. 2017 Jan;32(1):12-18. doi: 10.1111/jgh.13477. PMID 27349220